CLINICAL TRIAL: NCT04238429
Title: Efficacy of a Commercial Dentifrice Containing 10% High Cleaning Silica Base, 0.5% Sodium Phytate and 0.5% Sodium Pyrophosphate on Tooth Whitening: A 8-week Clinical Study in Adults in China
Brief Title: Whitening Efficacy of Dentifrice Containing 10% High Cleaning Silica, 0.5% Sodium Phytate and 0.5% Sodium Pyrophosphate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Liu Hongchun, Principal Investigator, Hospital of Stomatology, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Toothpaste whitenning
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Tooth Bleaching
Keywords: Toothpastes; Controlled Clinical Trial
MeSH Terms: interventions — Phytic Acid; sodium pyrophosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toothpaste containing effective ingredients (Experimental): Use the toothpaste containing 10% high cleaning silica base,0.5% sodium phytate and 0.5% sodium pyrophosphate to brush teeth twice daily for 8 weeks
  Interventions: Drug: Toothpaste containing 10% high cleaning silica base, 0.5% sodium phytate and 0.5% sodium pyrophosphate
- Negative control toothpaste (Placebo Comparator): Use the negative control dentifrice to brush teeth twice daily for 8 weeks
  Interventions: Drug: Control toothpaste

INTERVENTIONS:
Drug: Toothpaste containing 10% high cleaning silica base, 0.5% sodium phytate and 0.5% sodium pyrophosphate — Use the toothpaste to brush teeth twice a day for 8 weeks
  Arms: Toothpaste containing effective ingredients
Drug: Control toothpaste — Use the toothpaste to brush teeth twice a day for 8 weeks
  Arms: Negative control toothpaste

SUMMARY:
The objective of the present study was to compare the effects of a commercially available dentifrice containing 10% high cleaning silica base, 0.5% sodium phytate and 0.5% sodium pyrophosphate versus a negative control dentifrice on removal of extrinsic stains.

DETAILED DESCRIPTION:
There is great concern on the tooth esthetics and color among people, especially young adults. Great efforts have been made in order to improve patients' smile. Epidemiological studies have reported that dissatisfaction with tooth color ranged from 19.6% to 65.9%, depending on different population. An oral health related quality of life questionnaire for use among young adults reported that tooth color was the most important concern. This dissatisfaction with tooth color has been shown to be associated with increased desire for treatments that improve dental aesthetics including tooth whitening dentifrices. Tooth whitening products generally help to improve the overall whiteness of teeth, by removing and controlling the formation of extrinsic stains. In recent years the interest on the treatment of tooth stain with various tooth whitening agents, among which dentifrice containing high cleaning silica is widely used.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-70 years old
* Good general health
* Could attend the clinical examinations during the 8 week study period
* Possessing >20 natural permanent teeth that were uncrowned or heavily filled with restorative materials, excluding third molars
* Having a whole-mouth mean tooth stain score of more than 1.5 according to the Lobene index.

Exclusion Criteria:

* Severe oral diseases, chronic disease or allergic to the trial products
* Advanced periodontal diseases
* Females who are pregnant or lactating
* Taking part in other clinical trials
* Taking part in orthodontic treatment or wearing removable denture
* Fluorosis or tetracycline teeth
* Receiving prophylaxis during the previous 3 months or tooth whitening treatment during the past 6 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongchun Liu, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Guanghua School of Stomatology, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu H, Tu J. Reduction of extrinsic tooth stain by a toothpaste containing 10% high cleaning silica, 0.5% sodium phytate and 0.5% sodium pyrophosphate: an 8-week randomised clinical trial. BMC Oral Health. 2021 Mar 11;21(1):113. doi: 10.1186/s12903-021-01484-5. PMID 33706750

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste
Started | 43 | 43
Completed | 40 | 41
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (9.22) | 42.05 (10.19) | 42.27 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 23 | 19 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  Han | 40 | 41 | 81
Region of Enrollment [Number; unit: participants]
  China | 40 | 41 | 81
Lobene Stain Index: Area [Mean (Standard Deviation); unit: units on a scale] — Tooth stain of the anterior teeth were measured using the Lobene Stain Index. The index measures the area and intensity of extrinsic tooth stain on the facial and lingual surfaces of the lower anterior teeth and facial surfaces of the upper anterior teeth. The tooth surfaces were divided into two parts: body and gingival. For each part, the stain area was assessed using 0-3 scale. 0= No stain detected; 1= stain covering up to 1/3 of the region; 2= Stain covering >1/3 to 2/3 of the region; 3=Stain covering >2/3 of the region.
  units on a scale | 1.63 (0.49) | 1.59 (0.45) | 1.61 (0.47)
Lobene Stain Index: Intensity [Mean (Standard Deviation); unit: units on a scale] — Tooth stain of the anterior teeth were measured using the Lobene Stain Index. The index measures the area and intensity of extrinsic tooth stain on the facial and lingual surfaces of the lower anterior teeth and facial surfaces of the upper anterior teeth. The tooth surfaces were divided into two parts: body and gingival. For each part, the stain intensity was assessed using 0-3 scale. 0= No stain; 1=Light stain(yellow to light brown or gray); 2=Moderate stain(medium brown); 3=Heavy stain(dark brown to black).
  units on a scale | 1.69 (0.64) | 1.72 (0.59) | 1.7 (0.61)
Lobene Stain Index: Composite [Mean (Standard Deviation); unit: units on a scale] — Tooth stain of the anterior teeth were measured using the Lobene Stain Index. The tooth surfaces were divided into two parts: body and gingival. For each part, the stain area was assessed using 0-3 scale and the stain intensity was assessed using 0-3 scale. Lobene Stain Index: Composite for each part is the product of the stain area and intensity scores. The minimum score for Lobene Stain Index: Composite is 0 when both the stain area and intensity scores are 0. The maximum score for Lobene Stain Index: Composite is 9 when both the stain area and intensity scores are 3.
  units on a scale | 3.7 (1.65) | 3.72 (1.53) | 3.71 (1.58)

OUTCOME MEASURES:

1. Primary Outcome: Lobene Stain Index of Stain Extent Scores 4 Weeks After Dentifrice Use
Description: Tooth stain of the anterior teeth were measured using the Lobene Stain Index. The index measures the area and intensity of extrinsic tooth stain on the facial and lingual surfaces of the lower anterior teeth and facial surfaces of the upper anterior teeth. The tooth surfaces were divided into two parts: body and gingival. For each part, the stain intensity was assessed using 0-3 scale. 0= No stain; 1=Light stain(yellow to light brown or gray); 2=Moderate stain(medium brown); 3=Heavy stain(dark brown to black).
Time Frame: 4 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste
Number analyzed (Participants) | 40 | 41
score on a scale | 1.35 (0.6) | 1.64 (0.65)

2. Primary Outcome: Lobene Stain Index of Stain Area Scores 4 Weeks After Dentifrice Use
Description: Tooth stain of the anterior teeth were measured using the Lobene Stain Index. The index measures the area and intensity of extrinsic tooth stain on the facial and lingual surfaces of the lower anterior teeth and facial surfaces of the upper anterior teeth. The tooth surfaces were divided into two parts: body and gingival. For each part, the stain area was assessed using 0-3 scale. 0= No stain detected; 1= stain covering up to 1/3 of the region; 2= Stain covering >1/3 to 2/3 of the region; 3=Stain covering >2/3 of the region.
Time Frame: 4 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste
Number analyzed (Participants) | 40 | 41
score on a scale | 1.1 (0.44) | 1.32 (0.47)

3. Primary Outcome: Lobene Stain Index of Stain Composite Scores 4 Weeks After Dentifrice Use
Description: Tooth stain of the anterior teeth were measured using the Lobene Stain Index. The tooth surfaces were divided into two parts: body and gingival. For each part, the stain area was assessed using 0-3 scale and the stain intensity was assessed using 0-3 scale. Lobene Stain Index: Composite for each part is the product of the stain area and intensity scores. The minimum score for Lobene Stain Index: Composite is 0 when both the stain area and intensity scores are 0. The maximum score for Lobene Stain Index: Composite is 9 when both the stain area and intensity scores are 3.
Time Frame: 4 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste
Number analyzed (Participants) | 40 | 41
score on a scale | 2.39 (1.35) | 3.23 (1.6)

4. Primary Outcome: Lobene Stain Index of Stain Extent Scores 8 Weeks After Dentifrice Use
Description: as for outcome 1
Time Frame: 8 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste
Number analyzed (Participants) | 40 | 41
score on a scale | 0.98 (0.49) | 1.33 (0.68)

5. Primary Outcome: Lobene Stain Index of Stain Area Scores 8 Weeks After Dentifrice Use
Description: as for outcome 2
Time Frame: 8 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste
Number analyzed (Participants) | 40 | 41
score on a scale | 0.83 (0.36) | 1.12 (0.46)

6. Primary Outcome: Lobene Stain Index of Stain Composite Scores 8 Weeks After Dentifrice Use
Description: as for outcome 3
Time Frame: 8 weeks after dentifrice use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste
Number analyzed (Participants) | 40 | 41
score on a scale | 1.45 (0.78) | 2.5 (1.52)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Toothpaste Containing Effective Ingredients | Negative Control Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT04238429/Prot_SAP_001.pdf